CLINICAL TRIAL: NCT07170995
Title: A Randomized, Open-label, Controlled, Multicenter Phase III Study of SHR-8068 Combined With Adebrelimab and Platinum-based Chemotherapy Versus Tislelizumab Combined With Platinum-based Chemotherapy as First-line Treatment for Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Phase III Study of SHR-8068 Combined With Adebrelimab and Chemotherapy Versus Tislelizumab Combined With Chemotherapy in the Treatment of Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-8068-302
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum Compounds; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-8068，adebelizumab and platinum-based chemotherapy (Experimental)
  Interventions: Drug: SHR-8068，adebelizumab and platinum-based chemotherapy
- tislelizumab, and platinum-based chemotherapy (Active Comparator)
  Interventions: Drug: tislelizumab, and platinum-based chemotherapy

INTERVENTIONS:
Drug: SHR-8068，adebelizumab and platinum-based chemotherapy — SHR-8068，adebelizumab and platinum-based chemotherapy
  Arms: SHR-8068，adebelizumab and platinum-based chemotherapy
Drug: tislelizumab, and platinum-based chemotherapy — tislelizumab, and platinum-based chemotherapy
  Arms: tislelizumab, and platinum-based chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, multicenter Phase III clinical trial to evaluate the efficacy and safety of SHR-8068 combined with adebrelimab and platinum-based chemotherapy versus tislelizumab combined with platinum-based chemotherapy as first-line treatment for advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years old, no gender limitation.
3. Newly diagnosed histologically or cytologically confirmed, locally advanced or metastatic non-small cell lung cancer (NSCLC) that is treatment naive and not amenable to curative therapy including surgical resection or chemoradiation.
4. Confirmed tumor PD-L1 status prior to randomization.
5. Eastern Cooperative Oncology Group (ECOG) score: 0-1
6. With a life expectancy ≥ 3 months.
7. At least one measurable lesion according to RECIST v1.1.

Exclusion Criteria:

1. Have untreated central nervous system metastasis; or have meningeal metastasis or spinal cord compression;
2. Uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites;
3. Previous or co-existing malignancies；
4. Have Active or prior documented autoimmune or inflammatory disorders;
5. Active hepatitis B or hepatitis C, or with a history of immunodeficiency;
6. Have an active or past medical history of interstitial lung disease (ILD)/pneumonitis, including drug-induced or radiation ILD/pneumonitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by Blinded Independent Central Review [BICR] | Approximately 32 months.
  PFS (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]) by BICR was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression)
OS | Approximately 64 months.
  OS was defined as the time from the date of randomization until death due to any cause.

SECONDARY OUTCOMES:
PFS by the investigator | Approximately 32 months.
  PFS (per RECIST 1.1) by the investigator was defined as time from date of randomization until date of objective disease or death (by any cause in the absence of progression)
Objective Response Rate (ORR) | Approximately 32 months.
  ORR (per RECIST 1.1) by BICR or the investigator was defined as the percentage of patients with at least one visit response of complete response (CR) or partial response (PR).
Duration of Response (DoR) | Approximately 32 month
  DoR (per RECIST 1.1) by BICR or the investigator was defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression.
Incidence and Severity of Adverse Events (AEs) | Approximately 64 months.
  Incidence and severity of treatment emergent adverse events (TEAEs) will be reported. Any adverse event occurring at or after the initial administration of study treatment through the day of last dose plus 60 days, or until the start of subsequent anticancer therapy (if earlier), is considered to be treatment emergent.
Time to Deterioration of PRO Symptoms, Assessed Using EORTC QLQ C30-Lung Cancer Module 13 (QLQ-LC13) | Approximately 64 months.
  The EORTC QLQ-LC13 is a disease-specific 13-item self-administered questionnaire for lung cancer, to be used in conjunction with the EORTC QLQ-C30. It comprises both multi-item and single-item measures of lung cancer-associated symptoms and treatment-related symptoms from conventional chemotherapy and radiotherapy. Scores from 0 to 100 were derived for each symptom item, with higher scores representing greater level of symptoms. Time to deterioration was defined as time from randomization until the date of first clinically meaningful deterioration that was confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided